CLINICAL TRIAL: NCT06304402
Title: Comparison of the Effects of Shoulder Stretching Exercise and Percussive Massage Treatment on Shoulder Rotation Movements and Attack Speed in Female Volleyball Players
Brief Title: Comparing Shoulder Stretching and Percussive Massage on Shoulder Rotation and Attack Speed in Female Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gonca Şahiner Pıçak, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7978-GOA
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation Stretching (Experimental): Proprioceptive Neuromuscular Facilitation Stretching Group participants will undergo one session of PNF posterior shoulder stretching exercise in the modified sleeper position.
  Interventions: Behavioral: The Proprioceptive Neuromuscular Facilitation Stretching
- The Percussive Massage Treatment (Experimental): The Percussive Massage Treatment Group participants will receive a 5-minute massage on the posterior deltoid area.
  Interventions: Device: The Percussive Massage Treatment

INTERVENTIONS:
Device: The Percussive Massage Treatment — In the group where regional vibration is applied, the Hypervolt™ vibrating massage device (HYPERICE Inc, US) will be used. This device is a vibration device with five different speed settings, vibrating at 3,200 percussions per minute (HYPERICE Inc. 'Hypervolt' device. Retrieved from https://hyperice.com/hypervolt-bluetooth, Accessed on: 08.12.2021). The device offers five different head attachment options. For this study, the ball attachment option will be selected as it is the least aggressive option, and the vibration from the device will be applied to the relevant muscle body (Kayoda, 2019). For facilitatory effect, the application will be performed on the posterior deltoid for 5 minutes at a low frequency.
  Arms: The Percussive Massage Treatment
Behavioral: The Proprioceptive Neuromuscular Facilitation Stretching — Among the PNF stretching techniques, the muscle-relaxation technique will be applied. The athlete will be positioned in a side-lying posture on the treatment table with the dominant shoulder in the modified sleeper position, ensuring stabilization of the scapula on the table. The other arm will be positioned in extension along the body with the palm facing upwards. The participant will be instructed to actively bring the arm of the lower limb to the physiological barrier of internal rotation. At this point, they will be asked to perform maximum isometric contraction in external rotation for 7 seconds. After the isometric contraction, the muscle will be relaxed, and active-assisted stretching will be applied in internal rotation for 15 seconds. A 5-second rest will be provided between repetitions, and the exercise will consist of 5 repetitions.
  Arms: Proprioceptive Neuromuscular Facilitation Stretching

SUMMARY:
This study aims to investigate the acute effects of PNF modified sleeper stretches and percussive massage treatment on shoulder rotation movements and attack speed in female volleyball players and compare these applications.

DETAILED DESCRIPTION:
56 female volleyball players will randomized into 2 groups of 28 people each. In the evaluations conducted on the participants, rotational normal joint movements of the athletes will be measured using a digital inclinometer. The spike velocities of the athletes will be determined using a sports radar (Sports Radar 3300, Sports Electronics Inc, Washington, D.C. USA.). Participants will be randomly divided into two different groups consisting of 28 individuals each. The Proprioceptive Neuromuscular Facilitation Stretching Group (PNFG) participants will undergo one session of PNF posterior shoulder stretching exercise in the modified sleeper position. The Percussive Massage Treatment Group (PMTG) participants will receive a 5-minute massage on the posterior deltoid area. Evaluations will be repeated three times before the applications, immediately after, and 30 minutes post-application and the effects of different applications will be compared through analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being a volleyball player
* Age between 14 and 40 years

Exclusion Criteria:

* Presence of shoulder pain
* History of fracture and surgery in the shoulder girdle
* Presence of systemic musculoskeletal disease
* Presence of glenohumeral instability (Positive apprehension, relocation, or subluxation test)
* Pain in the cervical region with upper extremity movements
* Experiencing shoulder problems requiring medical treatment within the last year

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Shoulder internal rotation range of motion | baseline measurements, 5 minutes and 30 minutes
  Change of shoulder internal rotation range of motion (with a digital inclinometer)

SECONDARY OUTCOMES:
Attack Speed | baseline measurements, 5 minutes and 30 minutes
  Change of attack speed of the volleyball players (with a radar gun)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yeşilyaprak, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No